CLINICAL TRIAL: NCT04805775
Title: Effect of Desflurane on Postoperative Sleep Quality in Patients Undergoing Elective Breast Surgery: A Non-inferiority Randomized Controlled Trial
Brief Title: Desflurane and Postoperative Sleep Quality in Patients Undergoing Elective Breast Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zhongnan Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: B076201420067
Record Dates: First submitted 2021-03-16; First posted 2021-03-18 (Actual); Last update posted 2023-05-31 (Actual); Status verified 2023-04

CONDITIONS: Desflurane; Propofol; Postoperative Sleep; PSQI; Breast Tumor
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Desflurane Inhalation Group (Experimental): Anesthesia maintenance: Desflurane inhalation (MAC 1.0-1.2) Sufentanil 0.3-0.5 μg / (kg·h) Cisatracurium 1-3 μg / (kg·min)
  Interventions: Drug: Desflurane Inhalation
- Propofol Group (Active Comparator): Anesthesia maintenance: Propofol TCI: 3-4ug / ml Sufentanil 0.3-0.5 μg / (kg·h) Cisatracurium 1-3 μg / (kg·min)
  Interventions: Drug: Desflurane Inhalation

INTERVENTIONS:
Drug: Desflurane Inhalation — Subjects were randomized in a 1:1 ratio to undergo breast surgery under maintenance of anesthesia with the classical intravenous anesthetic drug propofol (reference group) or the inhaled anesthetic drug desflurane (test group).

SUMMARY:
This study intends to investigate the effects of desflurane on postoperative sleep quality to guide perioperative patient management.

ELIGIBILITY:
Inclusion Criteria:

1. Undergoing elective breast surgery
2. Age 18-75 years old
3. ASA-PS grade I or II
4. Those who voluntarily participate in the research and sign the informed consent

Exclusion Criteria:

1. Cognitive impairment (MMSE <27) before the operation
2. The patients received adjuvant chemotherapy before the operation
3. At present, they are taking psychoactive, opioid, anti-anxiety, and hypnotic drugs
4. Known or treated patients with obstructive sleep apnea
5. Patients with other cancers

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2021-10-21 (Actual); Primary Completion 2022-09-09 (Actual); Study Completion 2023-03-10 (Actual)

PRIMARY OUTCOMES:
Pittsburgh sleep quality index | Postoperative 3rd day

SECONDARY OUTCOMES:
Pittsburgh sleep quality index | Postoperative 7th, and 30th days
Total sleep time (TST), Rapid eye movement time (REM), Wakefulness after sleep onset (WASO) | Postoperative 1st, 2nd, and 3rd days
  Fitbit Charge 2™ objectively measured
Self-Rating Anxiety Scale Scores | Postoperative 3rd, 7th, and 30th days
Self-Rating Depression Scale Scores | Postoperative 3rd, 7th and 30th days
Visual analogue scale scores | Postoperative 3rd, 7th and 30th days
Flurbiprofen dose | Postoperative 1st, 2nd, and 3rd days
Recovery time and quality (steward scores) | Up to 2 hours after operation

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongnan Hospital of Wuhan University, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wang X, Xiong B, Wu T, Liu X, Li K, Wang S, Deng MG, Peng M. Effect of desflurane maintenance on postoperative sleep quality in patients undergoing elective breast surgery: A non-inferiority randomized controlled trial. Sleep Med. 2024 Sep;121:287-294. doi: 10.1016/j.sleep.2024.07.022. Epub 2024 Jul 17. PMID 39038404